CLINICAL TRIAL: NCT01300260
Title: The Effect of LY2189265 on Insulin Secretion in Response to Intravenous Glucose Infusion
Brief Title: Effect of LY2189265 on Insulin Secretion in Response to Intravenous Glucose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 11371; H9X-MC-GBCI (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-02-03; First posted 2011-02-21 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Insulin; Insulin Lispro; Glucose; Glucagon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2189265 then Placebo (Experimental): LY2189265 (Dulaglutide) then Placebo: A single 1.5 milligram (mg) subcutaneous (SC) injection of LY2189265 on Day 1 in Period 1, followed by a single SC injection of Placebo on Day 1 in Period 2.
  On Day 3 of each period, participants underwent a 6-hour insulin infusion, followed by an intravenous (IV) dextrose bolus (0.3 gram/kilogram [g/kg] over approximately 2 minutes). Three hours later, participants were administered a second IV dextrose bolus of 25 g of 50% dextrose or a suitably adjusted dose according to glycemic status (20 g of 50% dextrose for participants with 3-hour glucose between 5.2 and 10 millimole/liter [mmol/L] or 15 g of 50% dextrose for participants with 3-hour glucose >10 mmol/L), followed by a 20% dextrose at the set infusion rate of 600 milliliter/hour [mL/h] for 35 minutes. Fifteen minutes after the start of the 20% dextrose infusion, an IV 1-mg glucagon bolus was administered.
  There was a washout period of at least 28 days between Periods 1 and 2.
  Interventions: Biological: LY2189265; Drug: Placebo; Drug: Insulin; Drug: Glucose; Drug: Glucagon
- Placebo then LY2189265 (Experimental): Placebo then LY2189265 (Dulaglutide): A single subcutaneous injection of Placebo on Day 1 in Period 1, followed by a single 1.5 milligrams (mg) subcutaneous injection of LY2189265 on Day 1 in Period 2.
  On Day 3 of each period, participants underwent a 6-hour insulin infusion, followed by an intravenous (IV) dextrose bolus (0.3 gram/kilogram [g/kg] over approximately 2 minutes). Three hours later, participants were administered a second IV dextrose bolus of 25 g of 50% dextrose or a suitably adjusted dose according to glycemic status (20 g of 50% dextrose for participants with 3-hour glucose between 5.2 and 10 millimole/liter [mmol/L] or 15 g of 50% dextrose for participants with 3-hour glucose >10 mmol/L), followed by a 20% dextrose at the set infusion rate of 600 milliliter/hour [mL/h] for 35 minutes. Fifteen minutes after the start of the 20% dextrose infusion, an IV 1-mg glucagon bolus was administered.
  There was a washout period of at least 28 days between Periods 1 and 2.
  Interventions: Biological: LY2189265; Drug: Placebo; Drug: Insulin; Drug: Glucose; Drug: Glucagon

INTERVENTIONS:
Biological: LY2189265 — Administered subcutaneously
  Other Names: Dulaglutide
Drug: Placebo — Administered subcutaneously
Drug: Insulin — Administered intravenously
  Other Names: Lispro
Drug: Glucose — Administered intravenously
  Other Names: Dextrose
Drug: Glucagon — Administered intravenously
  Other Names: Glucagon hydrochloride

SUMMARY:
The purpose of this study is to measure the effect of LY2189265 to increase insulin levels in response to glucose intake.

ELIGIBILITY:
Inclusion Criteria:

All Participants

* Women must be surgically sterile (hysterectomy or bilateral oophorectomy or tubal ligation) or postmenopausal as defined by age >45 years without use of oral contraceptive agents for greater than 1 year and have either:

  * spontaneous amenorrhea greater than 12 months, or
  * spontaneous amenorrhea 6 to 12 months with documented follicle stimulating hormone (FSH) >25 milli international units/milliliter (mIU/mL) and serum estradiol <73 picomoles/liter (pmol/L) (20 picograms/milliliter [pg/mL])
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the ethical review board governing the site
* Have serum creatinine <150 micromoles/liter (µmol/L) (<1.3 milligrams/deciliter [mg/dl] in women, <170 µmol/L [<1.5 mg/dL] in men)
* Have normal hemoglobin result, as determined by the investigator

Healthy Participants

* Overtly healthy men and women as determined by medical history, normal lab results and physical examination.
* Body mass index (BMI) between 19 and 25 kilograms/meter squared (kg/m^2), inclusive.
* Normal blood pressure and heart rate as determined by the investigator
* Have a normal response to an oral glucose tolerance test (OGTT) (glucose <7.8 millimoles/liter [mmol/L] [<140 mg/dL] at 2 hours after 75 grams (g) oral glucose load)

Participants with type 2 diabetes mellitus (T2DM)

* Participants will have a BMI between 22.0 and 40.0 kg/m^2
* Have T2DM controlled with diet and exercise alone or metformin for at least 4 weeks prior to admission
* Have a hemoglobin A1c (HbA1c) value at screening (or within 4 weeks prior to screening) of 6.0% to 9.5%
* Diagnosed with T2DM within the past 10 years
* Clinical laboratory test results within normal range or deemed clinically insignificant by the Investigator. Abnormalities of serum glucose, serum lipids, urinary glucose, and urinary protein consistent with T2DM are acceptable.
* Participants who are taking stable-dose prescription medications (for example, antihypertensive agents, aspirin, lipid-lowering agents) for treatment of concurrent medical conditions are permitted to participate providing the medication is not associated with development of torsade de pointes. However, use of beta-blockers and thiazide diuretics are not permitted during this study.

Exclusion Criteria:

All Participants

* Within 30 days of the initial dose of study drug, have received treatment with a drug that has not received regulatory approval for any indication
* Known allergies to Glucagon-Like Peptide 1 (GLP-1) related compounds
* Have previously completed or withdrawn from this study or any other study in the last year investigating glucagon-like peptides or incretin mimetics including exenatide (Byetta®)
* Regular use of known drugs of abuse and/or positive findings on urinary drug screening, other than findings consistent with medication prescribed by the participant's physician(s)
* History or presence of cardiovascular, respiratory, renal, endocrine (except T2DM), hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs or of constituting a risk when taking the study medication or interfering with the interpretation of data
* Have a history or presence of gastrointestinal disorder
* Poorly controlled hypertension (systolic greater than 160 millimeters of mercury [mmHg], diastolic greater than 95 mmHg) and/or evidence of labile blood pressure including symptomatic postural hypotension. Use of beta-blockers or thiazide diuretics is not permitted during the study
* Have a clinically significant history of cardiac disease or presence of active cardiac disease within 1 year of the screening period
* Evidence of hepatitis C and/or positive hepatitis C antibody
* Evidence of hepatitis B and/or positive hepatitis B surface antigen
* Evidence of human immunodeficiency virus (HIV) and/or positive for HIV antibodies
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females) or are unwilling to follow alcohol restrictions (1 unit = 12 ounces [oz] or 360 milliliters[mL] of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Smoke more than 10 cigarettes or equivalent in nicotine use or nicotine substitutes per day
* Regular use of systemic corticosteroids by oral, intravenous, or intramuscular route, or potent, inhaled, or intranasal steroids known to have a high rate of systemic absorption
* Have a history or presence of significant active neuropsychiatric disease
* Blood donation of more than 500 mL in the last 3 months or any blood donation within the last month
* Any other condition, which in the opinion of the investigator would preclude participation in the study
* An abnormality in the 12-lead electrocardiogram (ECG) that in the opinion of the investigator increases the risk of participating in the study.
* Any clinically significant abnormal hematology, clinical chemistry, or urinary result(s) as determined by the investigator
* Evidence of significant active uncontrolled endocrine or autoimmune abnormalities (for example thyroid disease, or pernicious anemia) as judged by the screening physician

Healthy Participants

* Intended use of over-the-counter or prescription medication 7 and 14 days, respectively, prior to dosing.

Participants with T2DM

* Clinically significant peripheral vascular occlusive disease (PVOD).
* Known severe exudative diabetic retinopathy
* Known significant autonomic neuropathy as evidenced by urinary retention, diabetic diarrhea, or gastroparesis
* Have experienced a ketoacidotic episode (pH less than 7.3) requiring hospitalization in the last 6 months
* Outpatient use of insulin for control of diabetes within the past 2 years
* Use of antidiabetic agents other than metformin in the 4 weeks prior to study entry or use of thiazolidinediones within 12 weeks of study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuss, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2189265 First, Then Placebo: Includes healthy participants or participants with T2DM. LY2189265 (Dulaglutide): Single 1.5 milligram (mg) subcutaneous (SC) injection on Day 1 of Period 1. Placebo: Single SC injection of Placebo on Day 1 of Period 2.
  On Day 3 of each period, participants received a 6-hour (hr) insulin infusion, followed by an intravenous (IV) dextrose bolus (50% dextrose bolus, 0.3 gram/kilogram [g/kg] over approximately 2 minutes [min]). Three hr later, a 2nd IV dextrose bolus 25 g of 50% dextrose or a suitably adjusted dose according to glycemic status (20 g of 50% dextrose for participants with 3-hr glucose between 5.2 and 10 millimole/liter [mmol/L] or 15 g of 50% dextrose for participants with 3-hr glucose >10 mmol/L) was administered, followed by a 20% dextrose at the set infusion rate of 600 milliliter/hr [mL/hr] for 35 min. Fifteen min after the start of the 20% dextrose infusion, an IV 1-mg glucagon bolus was administered.
  There was a washout period of ≥28 days between Periods 1 & 2.
- Placebo First, Then LY2189265: Includes healthy participants and participants with T2DM. Placebo: Single subcutaneous (SC) injection of Placebo on Day 1 of Period 1. LY2189265 (Dulaglutide): Single 1.5 milligram (mg) SC injection on Day 1 of Period 2.
  On Day 3 of each period, participants received a 6-hour (hr) insulin infusion, followed by an intravenous (IV) dextrose bolus (50% dextrose bolus, 0.3 gram/kilogram [g/kg] over approximately 2 minutes [min]). Three hr later, a 2nd IV dextrose bolus 25 g of 50% dextrose or a suitably adjusted dose according to glycemic status (20 g of 50% dextrose for participants with 3-hr glucose between 5.2 and 10 millimole/liter [mmol/L] or 15 g of 50% dextrose for participants with 3-hr glucose >10 mmol/L) was administered, followed by a 20% dextrose at the set infusion rate of 600 milliliter/hr [mL/hr] for 35 min. Fifteen min after the start of the 20% dextrose infusion, an IV 1-mg glucagon bolus was administered.
  There was a washout period of ≥28 days between Periods 1 & 2.
Period: Period 1 of Study: First Intervention
Arm/Group | LY2189265 First, Then Placebo | Placebo First, Then LY2189265
Started | 15 | 17
Received at Least 1 Dose of Study Drug | 15 | 17
Completed | 14 | 16
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout Period of at Least 28 Days
Arm/Group | LY2189265 First, Then Placebo | Placebo First, Then LY2189265
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0
Period: Period 2 of Study: Second Intervention
Arm/Group | LY2189265 First, Then Placebo | Placebo First, Then LY2189265
Started | 14 | 16
Completed | 14 | 15
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Healthy participants or participants with type 2 diabetes mellitus (T2DM) who received at least one dose of study drug (LY2189265 or Placebo).
Groups:
- Healthy Participants: Includes healthy participants randomized to receive 1.5 milligram (mg) LY2189265 (Dulaglutide) first or Placebo first on Day 1 of either treatment sequence.
- Participants With Type 2 Diabetes Mellitus (T2DM): Includes participants with T2DM randomized to receive 1.5 mg LY2189265 (Dulaglutide) first or Placebo first on Day 1 of either treatment sequence.
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Participants With Type 2 Diabetes Mellitus (T2DM) | Total
Number analyzed (Participants) | 10 | 22 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (5.0) | 56.3 (6.1) | 54.9 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 7 | 15 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 22 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 22 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 22 | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximum Insulin Concentration (Cmax) - First Phase Response
Description: On Day 1 of each treatment period, all participants (healthy or with type 2 diabetes mellitus [T2DM]) received a single subcutaneous dose of either LY2189265 or placebo. On Day 3 of each treatment period, participants underwent a 6-hour insulin infusion, followed by an intravenous (IV) dextrose 50% bolus to stimulate insulin secretion. Three hours later, participants were administered a second dextrose bolus, followed by an infusion of 20% dextrose and, 15 minutes after the start of the 20% dextrose infusion, a 1-mg glucagon bolus was administered. Maximum plasma insulin concentration from 0 to 10 minutes (INSCmax[0-10]) following the first dextrose bolus (the first phase response) was corrected for baseline, where baseline was the mean of the insulin concentrations obtained between -30 and 0 minutes relative to the first dextrose bolus.
Time Frame: 0-10 minutes after dextrose bolus on Day 3 postdose
Population: All participants (healthy and with type 2 diabetes mellitus [T2DM]) who received at least 1 dose of study drug (LY2189265 or Placebo) with evaluable INSCmax(0-10) first response phase data.
Measure: Geometric Mean (95% Confidence Interval); unit: picomole per liter (pmol/L)
Groups:
- Healthy Participants: Placebo: Healthy participants first received a single subcutaneous injection of Placebo on Day 1. On Day 3, participants received a 6-hour insulin infusion followed by a dextrose bolus (50% dextrose bolus, 0.3 gram/kilogram [g/kg] over approximately 2 minutes).
- Healthy Participants: LY2189265: Healthy participant first received a single subcutaneous injection of 1.5 milligram (mg) LY2189265 on Day 1. On Day 3, participants received a 6-hour insulin infusion followed by a dextrose bolus (50% dextrose bolus, 0.3 gram/kilogram [g/kg] over approximately 2 minutes).
- Participants With Type 2 Diabetes Mellitus (T2DM): Placebo: T2DM participants first received a single subcutaneous injection of Placebo on Day 1. On Day 3, participants received a 6-hour insulin infusion followed by a dextrose bolus (50% dextrose bolus, 0.3 gram/kilogram [g/kg] over approximately 2 minutes).
- Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265: T2DM participants first received a single subcutaneous injection of 1.5 milligram (mg) LY2189265 on Day 1. On Day 3, participants received a 6-hour insulin infusion followed by a dextrose bolus (50% dextrose bolus, 0.3 gram/kilogram [g/kg] over approximately 2 minutes).
Arm/Group | Healthy Participants: Placebo | Healthy Participants: LY2189265 | Participants With Type 2 Diabetes Mellitus (T2DM): Placebo | Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265
Number analyzed (Participants) | 10 | 10 | 21 | 20
picomole per liter (pmol/L) | 233 [154 to 352] | 689 [455 to 1041] | 74.3 [46.8 to 118] | 401 [252 to 637]
Statistical Analysis 1: Comparison: Healthy Participants: Placebo vs Healthy Participants: LY2189265; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is two-sided; The mixed model analysis included treatment, period, and sequence as fixed effects and participant nested in sequence as a random effect; Geometric least squares (LS) mean ratio = 2.96, 95% CI 2-sided [2.41 to 3.64]
Statistical Analysis 2: Comparison: Participants With Type 2 Diabetes Mellitus (T2DM): Placebo vs Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is two-sided; [statistical method as in outcome 1, analysis 1]; Geometric least squares (LS) means ratio = 5.40, 95% CI 2-sided [4.09 to 7.13]

2. Primary Outcome: Area Under the Insulin Concentration-time Curve (AUC) - First Phase Response
Description: On Day 1 of each treatment period, all participants (healthy or with type 2 diabetes mellitus [T2DM]) received a single subcutaneous dose of either LY2189265 or placebo. On Day 3 of each treatment period, participants underwent a 6-hour insulin infusion, followed by an intravenous (IV) dextrose 50% bolus to stimulate insulin secretion. Three hours later, participants were administered a second dextrose bolus, followed by an infusion of 20% dextrose and, 15 minutes after the start of the 20% dextrose infusion, a 1-mg glucagon bolus was administered. Area under the plasma insulin concentration time curve from 0 to 10 minutes (INSAUC[0-10]) following the first dextrose bolus (the first phase response) was corrected for baseline, where baseline was the mean of the insulin concentrations obtained between -30 and 0 minutes relative to the first dextrose bolus.
Time Frame: 0-10 minutes after dextrose bolus on Day 3 postdose
Population: All participants (healthy and with type 2 diabetes mellitus [T2DM]) who received at least 1 dose of study drug (LY2189265 or Placebo) with evaluable INSAUC(0-10) first phase response data.
Measure: Geometric Mean (95% Confidence Interval); unit: picomole times hour per liter (pmol*h/L)
Arm/Group | Healthy Participants: Placebo | Healthy Participants: LY2189265 | Participants With Type 2 Diabetes Mellitus (T2DM): Placebo | Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265
Number analyzed (Participants) | 10 | 10 | 21 | 20
picomole times hour per liter (pmol*h/L) | 22.9 [15.0 to 34.9] | 70.7 [46.3 to 108] | 5.06 [2.90 to 8.83] | 40.1 [22.8 to 70.3]
Statistical Analysis 1: Comparison: Healthy Participants: Placebo vs Healthy Participants: LY2189265; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is two-sided; [statistical method as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 3.09, 95% CI 2-sided [2.66 to 3.59]
Statistical Analysis 2: Comparison: Participants With Type 2 Diabetes Mellitus (T2DM): Placebo vs Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is two-sided; [statistical method as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 7.92, 95% CI 2-sided [4.82 to 13.0]

3. Primary Outcome: Maximum Insulin Concentration (Cmax) - Second Phase Response
Description: On Day 1 of each treatment period, all participants (healthy or with type 2 diabetes mellitus [T2DM]) received a single subcutaneous dose of either LY2189265 or placebo. On Day 3 of each treatment period, participants underwent a 6-hour insulin infusion, followed by an intravenous (IV) dextrose 50% bolus to stimulate insulin secretion. Three hours later, participants were administered a second dextrose bolus, followed by an infusion of 20% dextrose and, 15 minutes after the start of the 20% dextrose infusion, a 1-mg glucagon bolus was administered. Maximum plasma insulin concentration from 10 to 180 minutes (INSCmax[10-180]) following the first dextrose bolus (the second phase response) was corrected for baseline, where baseline was the mean of the insulin concentrations obtained between -30 and 0 minutes relative to the first dextrose bolus.
Time Frame: 10-180 minutes after dextrose bolus on Day 3 postdose
Population: All participants (healthy and with type 2 diabetes mellitus [T2DM]) who received at least 1 dose of study drug (LY2189265 or Placebo) with evaluable INSCmax(10-180) second response phase data.
Measure: Geometric Mean (95% Confidence Interval); unit: picomole per liter (pmol/L)]
Arm/Group | Healthy Participants: Placebo | Healthy Participants: LY2189265 | Participants With Type 2 Diabetes Mellitus (T2DM): Placebo | Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265
Number analyzed (Participants) | 8 | 8 | 21 | 20
picomole per liter (pmol/L)] | 89.2 [64.7 to 123] | 370 [269 to 511] | 95.9 [66.3 to 139] | 363 [250 to 526]
Statistical Analysis 1: Comparison: Healthy Participants: Placebo vs Healthy Participants: LY2189265; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is two-sided; [statistical method as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 4.15, 95% CI 2-sided [3.45 to 5.00]
Statistical Analysis 2: Comparison: Participants With Type 2 Diabetes Mellitus (T2DM): Placebo vs Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is two-sided; [statistical method as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 3.78, 95% CI 2-sided [2.99 to 4.78]

4. Primary Outcome: Insulin Area Under the Curve (AUC) - Second Phase Response
Description: On Day 1 of each treatment period, all participants (healthy or with type 2 diabetes mellitus [T2DM]) received a single subcutaneous dose of either LY2189265 or placebo. On Day 3 of each treatment period, participants underwent a 6-hour insulin infusion, followed by an intravenous (IV) dextrose 50% bolus to stimulate insulin secretion. Three hours later, participants were administered a second dextrose bolus, followed by an infusion of 20% dextrose and, 15 minutes after the start of the 20% dextrose infusion, a 1-mg glucagon bolus was administered. Area under the plasma insulin concentration time curve from 10 to 180 minutes (INSAUC[10-180]) following the first dextrose bolus (the second phase response) was corrected for baseline, where baseline was the mean of the insulin concentrations obtained between -30 and 0 minutes relative to the first dextrose bolus.
Time Frame: 10-180 minutes after dextrose bolus on Day 3 post dose
Population: All participants (healthy and with type 2 diabetes mellitus [T2DM]) who received at least 1 dose of study drug (LY2189265 or Placebo) with evaluable INSAUC(10-180) second response phase data.
Measure: Geometric Mean (95% Confidence Interval); unit: picomole times hour per liter (pmol*h/L)
Arm/Group | Healthy Participants: Placebo | Healthy Participants: LY2189265 | Participants With Type 2 Diabetes Mellitus (T2DM): Placebo | Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265
Number analyzed (Participants) | 8 | 8 | 21 | 20
picomole times hour per liter (pmol*h/L) | 68.8 [41.7 to 114] | 141 [85.3 to 232] | 147 [103 to 209] | 357 [250 to 511]
Statistical Analysis 1: Comparison: Healthy Participants: Placebo vs Healthy Participants: LY2189265; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — P-value is two-sided; [statistical method as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 2.04, 95% CI 2-sided [1.26 to 3.31]
Statistical Analysis 2: Comparison: Participants With Type 2 Diabetes Mellitus (T2DM): Placebo vs Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is two-sided; [statistical method as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 2.44, 95% CI 2-sided [1.71 to 3.47]

5. Secondary Outcome: Insulin Maximum Concentration (Cmax)
Description: On Day 1 of each treatment period, all participants (healthy or with type 2 diabetes mellitus [T2DM]) received a single subcutaneous dose of either LY2189265 or placebo. Maximum plasma insulin concentration from -2 to 20 minutes following the glucagon bolus (INSCmaxG) is presented.
Time Frame: After glucagon bolus on Day 3 postdose
Population: All participants (healthy or with type 2 diabetes mellitus [T2DM]) who received at least 1 dose of study drug (LY2189265 or Placebo) with evaluable INSCmaxG data.
Measure: Geometric Mean (95% Confidence Interval); unit: picomole per liter (pmol/L)
Groups:
- Healthy Participants: Placebo: Healthy participants first received a single subcutaneous injection of Placebo on Day 1. On Day 3, participants received a 6-hour insulin infusion followed by a dextrose bolus 25 g of 50% dextrose or a suitably adjusted dose according to glycemic status (50% dextrose bolus, 0.3 gram/kilogram [g/kg] over approximately 2 minutes). Three hours later, participants were administered a second IV dextrose bolus 25 g of 50% dextrose or a suitably adjusted dose according to glycemic status (20 g of 50% dextrose for participants with 3-hour glucose between 5.2 and 10 millimole/liter [mmol/L] or 15 g of 50% dextrose for participants with 3-hour glucose >10 mmol/L), followed immediately by a 20% dextrose at the set infusion rate of 600 milliliter/hour [mL/h] for 35 minutes. Fifteen minutes after the start of the 20% dextrose infusion, an IV 1-mg glucagon bolus was administered.
- Healthy Participants: LY2189265: Healthy participants first received a single subcutaneous injection of Placebo on Day 1. On Day 3, participants received a 6-hour insulin infusion followed by a dextrose bolus (50% dextrose bolus, 0.3 gram/kilogram [g/kg] over approximately 2 minutes). Three hours later, participants were administered a second IV dextrose bolus 25 g of 50% dextrose or a suitably adjusted dose according to glycemic status (20 g of 50% dextrose for participants with 3-hour glucose between 5.2 and 10 millimole/liter [mmol/L] or 15 g of 50% dextrose for participants with 3-hour glucose >10 mmol/L), followed immediately by a 20% dextrose at the set infusion rate of 600 milliliter/hour [mL/h] for 35 minutes. Fifteen minutes after the start of the 20% dextrose infusion, an IV 1-mg glucagon bolus was administered.
- Participants With Type 2 Diabetes Mellitus (T2DM): Placebo: T2DM participants first received a single subcutaneous injection of Placebo on Day 1. On Day 3, participants received a 6-hour insulin infusion followed by a dextrose bolus (50% dextrose bolus, 0.3 gram/kilogram [g/kg] over approximately 2 minutes). Three hours later, participants were administered a second IV dextrose bolus 25 g of 50% dextrose or a suitably adjusted dose according to glycemic status (20 g of 50% dextrose for participants with 3-hour glucose between 5.2 and 10 millimole/liter [mmol/L] or 15 g of 50% dextrose for participants with 3-hour glucose >10 mmol/L), followed immediately by a 20% dextrose at the set infusion rate of 600 milliliter/hour [mL/h] for 35 minutes. Fifteen minutes after the start of the 20% dextrose infusion, an IV 1-mg glucagon bolus was administered.
- Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265: T2DM participants first received a single subcutaneous injection of 1.5 milligram (mg) LY2189265 on Day 1. On Day 3, participants received a 6-hour insulin infusion followed by a dextrose bolus (50% dextrose bolus, 0.3 gram/kilogram [g/kg] over approximately 2 minutes). Three hours later, participants were administered a second IV dextrose bolus 25 g of 50% dextrose or a suitably adjusted dose according to glycemic status (20 g of 50% dextrose for participants with 3-hour glucose between 5.2 and 10 millimole/liter [mmol/L] or 15 g of 50% dextrose for participants with 3-hour glucose >10 mmol/L), followed immediately by a 20% dextrose at the set infusion rate of 600 milliliter/hour [mL/h] for 35 minutes. Fifteen minutes after the start of the 20% dextrose infusion, an IV 1-mg glucagon bolus was administered.
Arm/Group | Healthy Participants: Placebo | Healthy Participants: LY2189265 | Participants With Type 2 Diabetes Mellitus (T2DM): Placebo | Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265
Number analyzed (Participants) | 8 | 8 | 20 | 20
picomole per liter (pmol/L) | 996 [716 to 1386] | 1215 [874 to 1690] | 1088 [827 to 1431] | 1514 [1151 to 1991]
Statistical Analysis 1: Comparison: Healthy Participants: Placebo vs Healthy Participants: LY2189265; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis — P-value is two-sided; [statistical method as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 1.22, 95% CI 2-sided [1.04 to 1.43]
Statistical Analysis 2: Comparison: Participants With Type 2 Diabetes Mellitus (T2DM): Placebo vs Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is two-sided; [statistical method as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 1.39, 95% CI 2-sided [1.27 to 1.53]

6. Other Pre Specified Outcome: Area Under the Insulin Concentration-time Curve (AUC)
Description: On Day 1 of each treatment period, all participants (healthy or with type 2 diabetes mellitus [T2DM]) received a single subcutaneous dose of either LY2189265 or placebo. Area under the plasma insulin concentration-time curve from -2 to 20 minutes following the glucagon bolus (INSAUCG) is presented.
Time Frame: After glucagon bolus on Day 3 postdose
Population: All participants (healthy or with type 2 diabetes mellitus [T2DM]) who received at least 1 dose of study drug (LY2189265 or Placebo) with evaluable INSAUCG data.
Measure: Geometric Mean (95% Confidence Interval); unit: picomole times hour per liter (pmol*h/L)
Groups:
- Healthy Participants: Placebo: Healthy participants first received a single subcutaneous injection of Placebo on Day 1. On Day 3, participants received a 6-hour insulin infusion followed by a dextrose bolus (50% dextrose bolus, 0.3 gram/kilogram [g/kg] over approximately 2 minutes). Three hours later, participants were administered a second IV dextrose bolus 25 g of 50% dextrose or a suitably adjusted dose according to glycemic status (20 g of 50% dextrose for participants with 3-hour glucose between 5.2 and 10 millimole/liter [mmol/L] or 15 g of 50% dextrose for participants with 3-hour glucose >10 mmol/L), followed immediately by a 20% dextrose at the set infusion rate of 600 milliliter/hour [mL/h] for 35 minutes. Fifteen minutes after the start of the 20% dextrose infusion, an IV 1-mg glucagon bolus was administered
- Healthy Participants: LY2189265: Healthy participant first received a single subcutaneous injection of 1.5 milligram (mg) LY2189265 on Day 1. On Day 3, participants received a 6-hour insulin infusion followed by a dextrose bolus (50% dextrose bolus, 0.3 gram/kilogram [g/kg] over approximately 2 minutes). Three hours later, participants were administered a second IV dextrose bolus 25 g of 50% dextrose or a suitably adjusted dose according to glycemic status (20 g of 50% dextrose for participants with 3-hour glucose between 5.2 and 10 millimole/liter [mmol/L] or 15 g of 50% dextrose for participants with 3-hour glucose >10 mmol/L), followed immediately by a 20% dextrose at the set infusion rate of 600 milliliter/hour [mL/h] for 35 minutes. Fifteen minutes after the start of the 20% dextrose infusion, an IV 1-mg glucagon bolus was administered.
Arm/Group | Healthy Participants: Placebo | Healthy Participants: LY2189265 | Participants With Type 2 Diabetes Mellitus (T2DM): Placebo | Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265
Number analyzed (Participants) | 8 | 8 | 20 | 20
picomole times hour per liter (pmol*h/L) | 239 [167 to 340] | 341 [239 to 486] | 236 [177 to 316] | 414 [310 to 554]
Statistical Analysis 1: Comparison: Healthy Participants: Placebo vs Healthy Participants: LY2189265; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis — P-value is two-sided; [statistical method as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 1.43, 95% CI 2-sided [1.14 to 1.80]
Statistical Analysis 2: Comparison: Participants With Type 2 Diabetes Mellitus (T2DM): Placebo vs Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is 2-sided; [statistical method as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 1.75, 95% CI 2-sided [1.59 to 1.94]

ADVERSE EVENTS:
Groups:
- Healthy Participants: Placebo: Healthy participants who received at least 1 subcutaneous injection of Placebo
- Healthy Participants: LY2189265: Healthy participants who received at least 1 subcutaneous injection of 1.5 milligram (mg) LY2189265
- Participants With Type 2 Diabetes Mellitus (T2DM): Placebo: T2DM participants who received at least 1 subcutaneous injection of Placebo
- Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265: T2DM participants who received at least 1 subcutaneous injection of 1.5 milligram (mg) LY2189265
Arm/Group | Healthy Participants: Placebo | Healthy Participants: LY2189265 | Participants With Type 2 Diabetes Mellitus (T2DM): Placebo | Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 2/10 | 6/10 | 9/21 | 11/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants: Placebo (N=10) | Healthy Participants: LY2189265 (N=10) | Participants With Type 2 Diabetes Mellitus (T2DM): Placebo (N=21) | Participants With Type 2 Diabetes Mellitus (T2DM): LY2189265 (N=21)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Infusion site phlebitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site phlebitis (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Injection site thrombosis (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days